CLINICAL TRIAL: NCT00660790
Title: Multifactorial Treatment of Cardiovascular Risk in Patients With Diabetes Mellitus Type-2: Identification of Treatment Non-Responders (The CARDIONOR Study)
Brief Title: Multifactorial Treatment of Cardiovascular Risk in Diabetic Patients: Identification of Treatment Non-Responders
Acronym: CARDIONOR
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Harald Sourij, MD, MD, Medical University of Graz
Other Study IDs: TCW 02/07
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type II
Keywords: diabetes mellitus type II, therapy non-responders
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes: diabetic subjects, above targets
  Interventions: Other: Intensified Treatment of risk factors

INTERVENTIONS:
Other: Intensified Treatment of risk factors — Patients received a target oriented, intensified treatment of risk factors according to current national treatment guidelines

SUMMARY:
The aim of the study is to develop a model that allows early identification of type-2 diabetic patients who will face progressive atherosclerosis despite intensive, multifactorial, target oriented treatment

DETAILED DESCRIPTION:
Background: Patients with type-2 diabetes face a substantially elevated risk for cardiovascular and cerebrovascular disease. This risk is based on traditional and non-traditional cardiovascular risk factors. It is, thus, partially mediated by modifiable conditions for instance blood pressure, cholesterol, or hyperglycemia. Indeed, controlled prospective intervention studies highlighted that individual lowering of those risk factors resulted in a reduction of vascular events such as acute coronary syndromes or stroke. The STENO-2 trial convincingly proved that multifactorial risk intervention, targeting all those risk factors substantially slowed the progression of atherosclerosis. As a result an even greater than 50 % reduction of vascular risk in patients with type-2 diabetes was observed. Thus, state of the art treatment for type-2 diabetic patients is multifactorial risk intervention targeting glucose control, lipids, blood pressure, platelets and the rennin-angiotensin-system.

Rationale: Risk normalisation for type-2 diabetic patients was not reached in the STENO-2 trial. In addition, it is, up to now, not possible to predict at early treatment stages who was to suffer progressive atherosclerosis and a future event despite intensive treatment of risk factors. Such early identification of treatment non-responders could enable to further intensify treatment or to develop new treatment strategies.

Aim: To develop a model that allows early identification of type-2 diabetic patients who will face progressive atherosclerosis despite intensive, multifactorial, target oriented treatment.

Experimental approach: To pursue the above mentioned aim, it will be investigated if, in patients with an indication to multifactorial risk intervention, either baseline characteristics or treatment responses after 3 months of intensified, multifactorial risk intervention can be used to predict progressive atherosclerosis during the study period of 2 years. To construct the model, traditional and non-traditional vascular risk factors will be evaluated.

Traditional vascular risk factors:

Traditional vascular risk factors may be grouped according to whether they may be modified or not. The major modifiable risk factors are hypertension, lipids, and hyperglycemia. All of them can be treated by lifestyle modification and pharmacologically. Smoking behaviour, sedentary lifestyle, nutrition and weight on the other hand may be influenced by lifestyle advice. Classic risk models such as the Framingham algorithm or the Prospective Cardiovascular Munster Study (PROCAM) model are based on traditional risk factors for risk estimation. They are, however, of limited applicability for diabetic patients due to the small number of such patients included and the lack of diabetes-specific variables in the model. From UK Prospective Diabetes Study (UKPDS) data a risk model for type-2 diabetes has been developed that describes future vascular risk based on such traditional risk factors including glycemic control and duration of diabetes. It is the only risk engine developed for a diabetic population. This model, however, does not take into account lipid lowering treatment in general, nor treatment responses to intensified intervention, nor novel vascular risk factors.

Novel, non-traditional vascular risk factors:

Endothelial dysfunction as well as inflammatory activity, reduced endothelial progenitor cells, and increased endothelial microparticles can be seen as more integral vascular risk factors or indicators, representing the combined influence of different traditional risk factors as well as specific vascular susceptibility. As such, they have been shown to be influenced by hyperglycemia, blood pressure or cholesterol. Specific treatment of those risk factors results in improvement of endothelial dysfunction, reduction of inflammatory activity, and increased number of endothelial progenitor cells.

Very recently, data from the Hoorn-study indicated that indeed about 43% of the excess vascular risk observed in diabetic patients is based on endothelial dysfunction and inflammatory activity. These data further point to the importance of non-traditional risk factors in the development of atherosclerosis and vascular events.

Progression of carotid artery intima media thickness (IMT) as a vascular endpoint:

The intima-media-thickness of the carotid arteries (IMT) is closely related to atherosclerotic burden in the coronary arteries and the risk for acute vascular events. It progressively increases over time, driven by age and cardiovascular risk factors. A high progression rate of IMT is indicative for future vascular events and treatment of risk factors reduces progression of IMT. Consequently, progression of IMT is a highly valid surrogate endpoint for progression of atherosclerosis and future vascular events.

Risk factors tested: Traditional risk factors:

Age, Gender, smoking behaviour, family history for coronary artery disease (CAD) or stroke, physical activity, lipids (total cholesterol, LDL-C, HDL-C, Triglycerides (TG), ApoA1, Apolipoprotein B (ApoB), Apo(a)), office blood pressure, serum creatinine, albuminuria, left ventricular hypertrophy (ECG)

Diabetes specific risk factors:

Duration of diabetes, HbA1c, fasting insulin, fasting proinsulin, fasting glycemia, Homeostasis Model Assessment (HOMA), glucose tolerance, BMI, waist circumference

Non-traditional risk factors:

Carotid artery IMT, prevalence and extend of carotid plaque, pulse wave velocity, vascular stiffness, ankle-brachial-index, endothelial function, inflammatory activity (both according to the Hoorn Study methods), endothelial progenitor cells, endothelial microparticles, plasminogen-activator-inhibitor-1 (PAI-1), tissue factor (TF).

Indication for multifactorial risk intervention: Based on the present knowledge type-2 diabetic patients are high risk subjects for the development of vascular disease and events. The excess risk, depending on the population studied is in the range of 2-6 fold. For that reason, every patient with type-2 diabetes per se has an indication for multifactorial risk intervention.

Intervention: Target oriented treatment of risk factors according to current treatment guidelines. Pharmacological therapy will be either newly installed or changed according the outline below.

All patients will receive comprehensive lifestyle counseling, personalized nutrition, and exercise advice.

After 3 months all modifiable or potentially variable risk factors will be evaluated again.

18 months after inclusion into the study carotid artery IMT will be measured again.

Outcome variables: The progression of IMT from baseline to 18 months will be the primary (dependent) outcome variable for the development of the model.

Modeling process: All risk factor variables to be tested for the model will be tested in univariate regression analyses with the progression of IMT as dependent variable. All variables with a p value below 0.200 will further be included into a multivariate regression analysis using a stepwise inclusion process.

Potential benefit: Early identification of type-2 diabetic patients who, despite intensified multifactorial risk intervention, face progressive atherosclerosis. Such patients, as a consequence could receive more individualized treatment by means of even more intensive intervention or application of different treatment strategies. As a result improved prevention of vascular events in type-2 diabetic patients could be finally reached.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type-2
* Indication to multifactorial risk intervention not in treatment target by means of two out of the following criteria:

  * Low Density Lipoprotein (LDL)-cholesterol > 120 mg/dl treated or untreated
  * Blood pressure: systolic >140 mmHg or diastolic >90 mmHg (office reading, treated or untreated)
  * (Glycated Hemoglobin) HbA1c > 7.5 % treated or untreated
* Signed informed consent
* Age 45 to 75 years
* Body Mass Index (BMI) < 35 kg/m2

Exclusion Criteria:

* History of any vascular event except angiography
* Heart failure > New York Heart Association (NYHA) II
* Serum Creatinine > 3.0 mg/dl
* Triglycerides > 400 mg/dl
* Aspartat-Aminotransferase (AST) / Alanin aminotransferase (ALT) > 3x Upper Limit of Normal (ULN)
* Major psychiatric disorder

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 Type-2 diabetic patients with no history of vascular events and need for therapy intensification.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Department of Internal Medicine, Medical University of Graz, Austria
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Result] Tripolt NJ, Meinitzer A, Eder M, Wascher TC, Pieber TR, Sourij H. Multifactorial risk factor intervention in patients with Type 2 diabetes improves arginine bioavailability ratios. Diabet Med. 2012 Oct;29(10):e365-8. doi: 10.1111/j.1464-5491.2012.03743.x. PMID 22803961
- [Result] Tripolt NJ, Narath SH, Eder M, Pieber TR, Wascher TC, Sourij H. Multiple risk factor intervention reduces carotid atherosclerosis in patients with type 2 diabetes. Cardiovasc Diabetol. 2014 May 23;13:95. doi: 10.1186/1475-2840-13-95. PMID 24884694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the outpatient clinic from the University Hospital of Graz.
Pre-assignment Details: 111 subjects were screened for the study between April 2008 and May 2010. Study inclusion criteria were met by 97 patients who were enrolled in the study.
Period: Baseline to 3 Months
Arm/Group | Patients With Type 2 Diabetes
Started | 97
Completed | 94
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Period: 3 Months to 2 Years
Arm/Group | Patients With Type 2 Diabetes
Started | 94
Completed | 77
Not Completed | 17
Not completed — Withdrawal by Subject | 17

BASELINE CHARACTERISTICS:
Groups:
- Patients With Type 2 Diabetes: patients with type 2 diabetes
  Intensified Treatment of risk factors: Patients received a target oriented, intensified treatment of risk factors according to current national treatment guidelines
Arm/Group | Patients With Type 2 Diabetes
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 97
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 91 (15)
Blood Pressure systolic [Mean (Standard Deviation); unit: mmHg] | 154 (17)
Blood Pressure diastolic [Mean (Standard Deviation); unit: mmHg] | 90 (9)
HbA1c (glycated hemoglobin) [Mean (Standard Deviation); unit: mmol/mol] | 66 (12)

OUTCOME MEASURES:

1. Primary Outcome: Change of Intima Media Thickness (IMT)
Description: Change of IMT from Baseline to 24 months
Time Frame: 24 months (from Baseline Visit to Visit 24 months after Baseline)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With Type 2 Diabetes
Number analyzed (Participants) | 77
mm | -0.023 (0.010)
Statistical Analysis 1: Comparison: Patients With Type 2 Diabetes; The paired student's t-test or the Wilcoxon signed-rank test was used to compare the measurements before and after multifactorial treatment, as appropriate, depending on the distribution of the data; Test type: Other; p = 0.021, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to study end (after 2 years).
Arm/Group | Patients With Type 2 Diabetes
All-Cause Mortality (participants affected / at risk) | 1/97
Serious Adverse Events (participants affected / at risk) | 18/97
Other Adverse Events (participants affected / at risk) | 35/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Type 2 Diabetes (N=97)
Insult (Vascular disorders) | 1 (1)
Gall bladder removal (Surgical and medical procedures) | 1 (1)
Kidney cyst (Renal and urinary disorders) | 1 (1) — inpatient stay due to kidney cyst
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
switch to insulin therapy (Metabolism and nutrition disorders) | 1 (1) — inpatient stay due to switch to insulin therapy
Cardiac insufficiency (Cardiac disorders) | 1 (1)
Insertion of stents (Cardiac disorders) | 1 (1)
Adenoma (Gastrointestinal disorders) | 1 (1) — inpatient stay due to clarifying adenoma
eye surgery (Eye disorders) | 1 (1) — inpatient stay
Spinal canal surgery (Surgical and medical procedures) | 1 (1)
Kidney tumor (Renal and urinary disorders) | 1 (1)
Tenodvaginitis stenosans (Surgical and medical procedures) | 1 (1)
chronic gastritis (Gastrointestinal disorders) | 1 (1)
diabetic arterial disease (Vascular disorders) | 1 (1)
Endarterectomy (Vascular disorders) | 1 (1)
Umbilical hernia (Surgical and medical procedures) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
prepyloric ulcera (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Type 2 Diabetes (N=97)
Hypoglycaemic Event (Metabolism and nutrition disorders) | 7 (16)
Nausea (General disorders) | 20 (30)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes